CLINICAL TRIAL: NCT02214888
Title: A 12 Week Double-blind, Randomized, Placebo-controlled Trial to Investigate Efficacy, Safety and Pharmacokinetics of BIRB 796 BS Tablets at Doses of 50 and 70 mg Administered Twice a Day in Patients With Active Rheumatoid Arthritis Who Have Failed at Least One DMARD
Brief Title: Efficacy, Safety and Pharmacokinetics of BIRB 796 BS Tablets in Patients With Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1175.18
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — doramapimod

ARMS (3):
- BIRB 796 BS, low dose (Experimental)
  Interventions: Drug: BIRB 796 BS, low dose; Drug: Placebo
- BIRB 796 BS, high dose (Experimental)
  Interventions: Drug: BIRB 796 BS, high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIRB 796 BS, low dose
  Arms: BIRB 796 BS, low dose
Drug: BIRB 796 BS, high dose
  Arms: BIRB 796 BS, high dose
Drug: Placebo
  Arms: BIRB 796 BS, low dose; Placebo

SUMMARY:
Study to determine the efficacy (including American College of Rheumatology (ACR) 20 response rate), safety, and pharmacokinetics of BIRB 796 BS as monotherapy in patients with moderate to severe rheumatoid arthritis who have failed at least one disease modifying antirheumatic drug (DMARD)

ELIGIBILITY:
Inclusion Criteria:

* Male or female from 18 to 75 years of age
* Diagnosis of rheumatoid arthritis (RA) established according to ACR criteria and date of diagnosis > 6 months
* Patient belonging to functional class I, II, or III
* Failure of at least one DMARD due to lack of efficacy or tolerability
* 2 out of the 3 following RA activity criteria: If this criterion is not met at visit 1, the whole set of RA activity criteria can be repeated at visit 2 (Repeated screening)

  * documentation of ≥ 9 swollen joints in a 66 joint count
  * documentation of ≥ 9 tender joints in a 68 joint count
  * C-reactive protein (CRP) ≥ 1.5 mg/dl or erythrocyte sedimentation rate (ESR) ≥ 28 mm/hr (or equivalent of ≥ 24mm/hr according to Panchenkov method)
* Written informed consent in accordance with Good Clinical Practice (GCP) and local legislation given prior to any study procedures, including washout of prohibited medications
* Only for centres participating in the pharmacokinetic (PK) substudy: Written informed consent in accordance with GCP and local legislation for participation in the PK substudy. Refusal to participate in the PK substudy is not an exclusion criterion for participation in the trial

Exclusion Criteria:

* Inflammatory rheumatic disease other than RA
* Treatment failure to a tumor necrosis factor (TNF)-blocking agent. Treatment failure is defined as not achieving at least an ACR 20 response (e.g. in a clinical trial) or - in clinical practice - having the TNF-blocking agent discontinued due to ineffectiveness
* History of vasculitis (characterised by e.g. nail bed hemorrhages or infarcts, vasculitic purpura, ulcers or gangrene, multisensory neuropathy, vasculitic retinopathy or scleritis of eyes). Isolated rheumatoid nodules of the skin are not a criterion for exclusion
* Serologic evidence of active hepatitis B and/or C
* Known HIV-infection
* History of prior tuberculosis infection or suspicion of active infection at screening based on results of chest x-ray not older than 6 months
* History of cardiovascular, renal, neurologic, psychiatric, liver, gastrointestinal, immunologic or endocrine dysfunction if they are clinically significant. A clinically significant disease is defined as one which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
* Recent history of heart failure (i.e. three years or less) or myocardial infarction (i.e. one year or less) or patients with any cardiac arrhythmia requiring drug therapy
* History of malignant disease in the last 5 years or suspicion of active malignant disease except successfully treated squamous or basal cell carcinoma of the skin
* Screening ECG results outside of the reference range of clinical relevance including, but not limited to QTcB > 480 msec, PR interval > 240 msec, QRS interval > 110 msec according to central ECG evaluation
* Clinically significant abnormal baseline hematology, blood chemistry or urinalysis if the abnormality defines a disease listed as an exclusion criterion or any of the following specific laboratory abnormalities: If this criterion is not met at visit 1, the laboratory assessments can be selectively repeated at visit 2 (Repeated screening)

  * alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin greater than upper limit of normal (ULN)
  * alkaline phosphatase, creatinine or white blood cell count greater than 1.5 x ULN
* History of drug or alcohol abuse within the past two years or active drug or alcohol abuse, present alcohol intake more than three drinks per day
* Female of childbearing potential (not 6 months post- menopausal or surgically sterilized) not using an approved form of birth control (hormonal contraceptives, oral or injectable/implantable, intra-uterine device (IUD))
* Inability to comply with the protocol
* Previous enrolment in this trial or previous exposure to BIRB 796 BS in another trial
* Hypersensitivity to trial drug

To be assessed at visit 3 (Baseline):

* Pregnancy (to be excluded by serum and urine beta human chorion-gonadotropin (βHCG)-test in women of childbearing potential) or breast feeding
* Active vasculitis
* Active infection or serious infectious diseases resulting in hospitalisation or requiring systemic anti-infective therapy within the last 4 weeks
* DMARD treatment within the last 4 weeks
* Last dose given within the specified time period for one of the following compounds or drugs:

  * Infliximab (Remicade®): 3 months
  * Adalimumab (D2E7): 3 months
  * Leflunomide: 3 months. If cholestyramine has been given for 10 days : 4 weeks
  * Investigational agent: 5- fold of the respective plasma half life or 4 weeks, whichever is longer
* Treatment with systemic corticosteroids in a dose higher than 10 mg/day prednisone equivalent
* Change in treatment with nonsteroidal antiinflammatory drugs (NSAIDs) or systemic corticosteroids within the last 4 weeks
* Synovectomy, joint surgery, radio-/chemo synoviorthesis, adrenocorticotropic hormone (ACTH) or any steroid injections (intraarticular, intravenous or intramuscular) within the last 4 weeks
* Participation in another clinical trial within the last 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2003-05; Primary Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Number of responders according to the American College of Rheumatology (ACR) 20 criteria | after 12 weeks of treatment

SECONDARY OUTCOMES:
Absolute differences to baseline in tender joint count (TJC, 68 joint count) | up to 12 weeks
Absolute differences to baseline swollen joint count (SJC, 66 joint count) | up to 12 weeks
Absolute differences to baseline in patients assessment of pain on a visual analogue scale (VAS) | up to 12 weeks
Absolute differences to baseline in patients global assessment of disease activity (PADA) on a VAS | up to 12 weeks
Absolute differences to baseline in physicians global assessment of disease activity on a VAS | up to 12 weeks
Absolute differences to baseline in patient's assessment of physical function measured by a standardised Health Assessment Questionnaire (HAQ) | up to 12 weeks
Absolute differences to baseline in concentration of C-reactive protein (CRP) | up to 12 weeks
Absolute differences to baseline in erythrocyte sedimentation rate (ESR) | up to 12 weeks
Number of responders to ACR 50 | after 12 weeks of treatment
Number of responders to ACR 70 | after 12 weeks of treatment
Number of responders to European League against Rheumatism (EULAR) response criteria | after 12 weeks of treatment
Number of drop-outs due to lack of efficacy, according to final assessment of investigator | after 12 weeks of treatment
Number of patients with adverse Events (AE) | up to 12 weeks after first drug administration
Number of patients with clinically relevant changes in laboratory tests | up to 12 weeks after first drug administration
Number of patients with clinically relevant changes in electrocardiogram (ECG) | up to 12 weeks after first drug administration
Number of patients with clinically relevant changes in vital signs | up to 12 weeks after first drug administration
Number of withdrawals due to AEs | up to 12 weeks after first drug administration
Cmax,ss (Maximum measured concentration of the analyte in plasma at steady state) | up to 24 hours after last drug administration
AUC0-t,ss (area under the drug plasma concentration-time curve over a dosing interval (t) at steady state | up to 24 hours after last drug administration
Cpre (predose concentration of the analyte in Plasma) | up to 24 hours after last drug administration
Cmin,ss (Minimum measured concentration of the analyte in plasma at steady state) | up to 24 hours after last drug administration